CLINICAL TRIAL: NCT02765932
Title: The Effect of a Psychosensory Therapy on Post-Op Pain in Hip and Knee Surgery: A Randomized Study
Brief Title: The Effect of a Psychosensory Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-00712
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Joint Replacement Surgery
Keywords: Hip; Knee; replacement; surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Therapy (Active Comparator): Dummy Movements
  Interventions: Procedure: Dummy Movements
- Psychosensory Therapy (Experimental): Will involve touch technique, havening.
  Interventions: Procedure: Psychosensory Therapy

INTERVENTIONS:
Procedure: Dummy Movements — The placebo group will be asked to perform the same touch technique and count backwards from 50 while removing petals from a flower. Patients will also perform these techniques before rehab and sleep.
  Arms: Placebo Therapy
Procedure: Psychosensory Therapy — The research assistant will administer one of the several psychosensory touch techniques prior to surgery. This will involve the touching of upper arms, palms, and a visualization process. This will last no longer than 10 minutes. These techniques will also be performed by the patients prior to any rehab sessions and before going to sleep. The patients will be asked to perform these touch techniques with the eyes closed and imaging having no pain. The patients will also be asked to keep a record of all medications.
  Arms: Psychosensory Therapy

SUMMARY:
This is a prospective study looking at the impact of psychosensory therapy and how it can diminish pain and consumption of pain medications. The primary study objective is to evaluate the change in Visual Analogue Score (VAS) score assessing for pain from Baseline, every day of inpatient stay, 7 days after leaving hospital (via phone), and 3 months post-op(via phone) and to correlate the psychosensory therapy and overall use of pain medications/narcotics.

DETAILED DESCRIPTION:
The study will aim to enroll 50 subjects. 25 subjects will receive placebo therapy which will be dummy movements while the other 25 will receive psychosensory therapy. The treatment group will involve a touch technique called havening.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing joint replacement surgery (Hip and Knee Only)
* Patient is willing to participate in pre- and postoperative surveys

Exclusion Criteria:

* Patients who have undergone joint replacement surgeries
* History of Chronic Narcotic Use (more than 30mg morphine dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Change in pain from baseline using Visual Analogue Score (VAS) | Baseline and 7 Months
  Measures level of Pain pre and post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States